CLINICAL TRIAL: NCT02421250
Title: Comparison of Accuracy and Clinical Outcomes of a Continuous Noninvasive Hemoglobin Monitor in the Emergency Room Setting
Brief Title: Noninvasive Hemoglobin Monitor in the ER
Acronym: SpHb
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI terminated the study prior to enrolling any participants.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB15-0167
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Hemoglobin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radical-7 Non-invasive Hgb Monitor (Experimental): We use the Radical-7 Noninvasive Hgb Monitor device (provided by Masimo Corporation from Irvine USA) to measure hemoglobin levels in patients in the experimental group.
  Interventions: Device: Radical-7 Noninvasive Hgb Monitor
- Control (No Intervention): We will use standard-of-care for control group and not use the SpHb monitor.

INTERVENTIONS:
Device: Radical-7 Noninvasive Hgb Monitor
  Arms: Radical-7 Non-invasive Hgb Monitor

SUMMARY:
The study is a clinical trial to determine whether more efficient medical and operational outcomes can be achieved with using the new SpHb monitoring during triage in the emergency room setting. The investigators also evaluate the accuracy of the measurements of the SpHb device by Maximo versus the gold standard of central hospital laboratory value. In addition, the investigators will assess patient satisfaction with the tool.

DETAILED DESCRIPTION:
A major issue faced by emergency departments all over the world is overcrowding, resulting from limited resources (i.e. staff, space, equipment) attending to a large of patients that exceeds the physical and/or staffing capacity of the ED. To manage the issue of overcrowding, the system of triage was created to help prioritize each patient's case, based on set criteria to determine time to treatment and/or which treatment is indicated. Our study will contribute to the discovery of more efficient ways of triaging patients based on objective and subjective criteria for decision-making about treatment and disposition, while simultaneously maintaining patient safety.

The investigators achieve this aim by evaluating the efficiency of a noninvasive and continuous total hemoglobin (SpHb) monitor provided by Masimo Corporation (Irvine USA). Standard hemoglobin measurements via central laboratory testing are invasive, painful, time-consuming, have increased lag time for analysis, potentially expose health care workers to blood-borne illness, and delay treatment onset because they require direct blood sampling. The new SpHb monitor potentially offers a new way to evaluate objective criteria about patients to maximize treatment outcomes and appropriate dispositions. The SpHb monitor has the potential to trend hemoglobin monitoring, quicken the detection of acute anemia, and avoid the complications, anxiety, expense, and patient discomfort associated with invasive blood draws.

In the ED setting, there is a need to efficiently triage a patient and designate a disposition for appropriate treatment management and outcomes. Hemoglobin level is an accurate indicator that helps distinguish patients who need early blood transfusion and meet criteria for admission. Noninvasive technology, such as the SpHb device by Masimo, will assist with common goals in emergency medicine: to efficiently and accurately decrease wait times to treatment and disposition, screening patients who have difficult venous access, providing repeated sampling without causing iatrogenic blood loss linked to anemia, and offering an approach that may be used to develop an organized coherent therapeutic plan based on physiologic criteria for the emergency patient as he/she proceeds from the ED to the OR, the hospital general floor, and the ICU.

This study will be performed at the University of Chicago Medical Center in the main adult emergency room. Patients will be examined and enrolled into our study initially by the triage nurse after each person has given his/her written informed consent.

Randomization process will be carried out based on days of the week. Patients will be enrolled in one group every two days. For example, starting on the week when we begin the trial, we will assign Monday patients to the control group, Tuesday patients to the experimental group, Wednesday patients to the control group… Two groups are similar in characteristics. Depending on whether the subject has been randomized into the control or experimental group, we will not use or use the SpHb monitor to obtain measurements. To obtain measurements, we place the probe of the device on the patient's finger and record the hemoglobin level determined by the Masimo Radical-7 Pulse CO-Oximeter.

We will collect patient satisfaction data 2 minutes after the placement of the SpHb device and 2 minutes after the blood sampling. The collection of blood is considered standard of care. Along with recording hemoglobin measurements, we will record triage chief complaint, final physician diagnosis, time to blood products transfusion, time to disposition (i.e. discharge home or Hospital admission via intensive care unit or general floor), time to procedure (i.e. procedure via operating room, endoscopy with interventional gastroenterology, interventional pulmonology, or ENT, or interventional radiology), and hemodynamics (i.e. blood pressure, heart rate, oxygen saturation, and respiratory rate).

ELIGIBILITY:
Inclusion Criteria: The following is the inclusion criteria for each participant based on initial complaints in triage of bleeding:

* GI bleeding-melena, hematochezia, hematemesis
* Vaginal bleeding
* Epistaxis
* Hematuria
* Hemoptysis
* Sickle cell patients
* Bleeding from recent surgical procedure
* Dizziness or lightheadedness in LVAD patients or hematology and oncology patients (i.e. cancer, leukemia, lymphoma-currently receiving chemo, stem cell treatment, or bone marrow transplant).

Exclusion Criteria:

* Exclusion criteria would consist of those patients in critically ill condition i.e. trauma, those needing massive transfusion protocol, cardiac arrest with active CPR, active seizure, hypothermia, acute intoxication/AMS that prohibits cooperation or following commands

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin Measurements | During intervention period (8 weeks)
  Hemoglobin level to be measured once at triage; hgb measurements (g/dL)

SECONDARY OUTCOMES:
Time to procedure | During intervention period (8 weeks)
  Measured in minutes; i.e. procedure via operating room, endoscopy with interventional gastroenterology, interventional pulmonology, or ENT, or interventional radiology

OTHER OUTCOMES:
Time to disposition | During intervention period (8 weeks)
  Measured in minutes
Time to blood transfusion | During intervention period (8 weeks)
  Measured in minutes
Hemodynamics | During intervention period (8 weeks)
  i.e. blood pressure, heart rate, oxygen saturation, and respiratory rate
Triage chief complaint | During intervention period (8 weeks)
  Reason for visiting the ER
Final physician diagnosis | During intervention period (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spiegel, MD MBA, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States